CLINICAL TRIAL: NCT05012813
Title: Feasibility of Substitution of Volatile Organic Compound Humidification to Simulate the Forest Experience Effects on Immune System Recovery
Brief Title: Humidified Forest Oils for Immune System Recovery in Stage I-III Breast or Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Amy M. Ross Ph.D., Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00023183; NCI-2021-08489 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00023183 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2021-08-06; First posted 2021-08-19 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Breast Carcinoma; Prostate Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms | interventions — Aromatherapy; Oils, Volatile; Coal Tar; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (SFIT, biospecimen, interview) (Experimental): Patients participate in SFIT, using humidified wood and fragrance oils, over 1 hour. on day 1, day 3 or 4 and on day 7. Patients also undergo blood sample collection at baseline and on days 3 or 4 and 7 and participate in interviews at baseline and post-treatment.
  Interventions: Other: Aromatherapy with Essential Oils

INTERVENTIONS:
Other: Aromatherapy with Essential Oils — Participate in SFIT this is one intervention with aroma therapy with essential Forest oils
  Other Names: Therapeutic Interventions; Therapeutic Method; Therapeutic Procedure; Therapeutic Technique; Therapy

SUMMARY:
This clinical trial studies the feasibility of simulating forest therapy using humidified wood or fragrant oils, in improving immune cells, like natural killer cells, number and activity, and their downstream proteins, perforin and granulysin in patients with stage I-III breast or prostate cancer who completed chemo- and/or radiation therapy. The knowledge gained from this study may help cancer patients who have compromised immune systems and who also cannot participate in outdoor activities like exercise or forest walks.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the feasibility of using humidified phytoncides to simulate the forest greenspace immersion (simulated forest immersion therapy [SFIT]) in cancer patients with solid tumor who have completed surgery, chemo- and radiation therapy as an alternate method of access to the natural forest greenspace.

SECONDARY OBJECTIVE:

I. Determine the feasibility of collecting and analyzing immune system measures while deploying the simulated forest immersion therapy with forest oils (SFIT), as well as measuring natural killer (NK) cell number and activity, and perforin and granulysin.

OUTLINE:

Patients participate in SFIT, using humidified wood and fragrance oils, over 1 hour on day 1, day 3 or 4 and on day 7. Patients also undergo blood sample collection at baseline and on days 3 or 4 and 7 and participate in interviews at baseline and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years. Both men and women and members of all races and ethnic groups will be included
* Participants must have histologically or cytologically confirmed breast cancer or prostate cancer (hormone therapy excepted) who are in stage I-V with or without evidence of metastasis using the Cancer Therapy Evaluation Program (CTEP) Simplified Disease Classification
* Participants must be within 12 months of their first diagnosis of breast or prostate cancer
* Criteria for solid tumors: Participants must have measurable disease, per doctor of medicine (MD) and data in medical record
* Participants must have no history of autoimmune disease
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* If they have asthma. Rationale: forest oils may be a possible trigger for asthma
* If they have a known allergy to citrus peel or pine forests. Rationale: forest oils may cause contact dermatitis and coughing
* If they are unable to detect common odors from commercial fragrances. Rationale, forest oils are humidified as an aroma to be inhaled in the simulate the forest greenspace immersion (SFIT)
* First diagnosis of breast or prostate cancer is longer than 12 months ago. Rationale, NK cell number recovery may be complete by this time after first treatment
* Febrile illness/infection within previous two weeks. Rationale, immune biomarkers will reflect previous febrile illness
* Current tobacco or tobacco use within 1 hour of start of SFIT. Rationale: forest oils may cause contact dermatitis and coughing
* Prior autoimmune disease, are on immune-modulating therapies (endocrine therapy allowed). Rationale, because of their poor prognosis rather than being in early stages of cancer
* Had surgery or invasive procedure in the past two months. Rationale, because of their poor prognosis rather than being in early stages of cancer
* Inability to complete study requisites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Humidified phytoncides to simulate the forest greenspace immersion (SFIT) | Baseline/Day 1
  Feasibility analysis will include qualitative interview data blinded by participant, CRC/research assistant and principal investigator. Qualitative interview questions include ease of use/deployment of humidified forest oils by the CRC/research assistant and PI, the ability of the participants to tolerate SFIT. The responses will be coded, themed and summarized will be used to determine the feasibility of intervention deployment and creation of a standardized procedure for future research. To determine dose drop off between the start of SFIT and the end of SFIT of the humidified phytoncides a t-test with an alpha level of 0.05 will be used.

SECONDARY OUTCOMES:
Collecting and analyzing immune system measures while deploying the simulated forest immersion therapy with forest oils | Baseline and at day 3 or 4 and on Day 7
  Will measure natural killer (NK) cell number and activity, and perforin and granulysin. NK cell number (NK CD3-/CD56+/) and activity (NK CD3-/CD56+/CD69+) will be tested with Flow Cytology. Perforin and granulysin will be tested by ELISA. Will use a t-test to determine the differences between these 4 variables collected at baseline and a Day 3-4. An alpha level of 0.05 will be set. Alternate analysis, the change NK cell number and activity will be determined from the mean of the standard range.

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Ross, Ph.D., Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided